CLINICAL TRIAL: NCT00773669
Title: Male Breast Cancer Summa Health System/Akron City Hospital Experience 1995-2007
Status: Completed | Type: Observational
Sponsor: Summa Health System (Other)
Responsible Party: Sponsor
Other Study IDs: Male Breast Cancer
Record Dates: First submitted 2008-10-15; First posted 2008-10-16 (Estimated); Last update posted 2013-05-31 (Estimated); Status verified 2013-05

CONDITIONS: Breast Cancer
Keywords: male breast cancer; Male breast cancer patients diagnosed and/or; treated at Summa Health System/Akron City Hospital; from the reference year of 1995 through 2007.
MeSH Terms: conditions — Breast Neoplasms; Breast Neoplasms, Male

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The primary goal of this retrospective study is to evaluate the male breast cancer patient population at Summa Health System/Akron City Hospital over a period of 18 years and compare the findings to historical data.

The objectives are to:

* identify risk factors.
* evaluate stage and histology at the time of presentation.
* document treatment modalities and outcomes.
* analyze outcomes for comparison to historical data.

ELIGIBILITY:
Inclusion Criteria:

* Male breast cancer patients diagnosed and/or treated at Summa Health System/Akron City Hospital from the reference year of 1995 through 2007.

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Males with breast cancer.
Sampling Method: Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2008-10; Primary Completion 2011-03 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Retrospective chart review to evaluate the male breast cancer patient population at Summa Health System/Akron City Hospital over a period of years and compare the findings to historical data. | Chart review from 1995-2007

CONTACTS AND LOCATIONS:
Overall Officials: Gary Williams, MD, Principal Investigator — Summa Health System